CLINICAL TRIAL: NCT03703726
Title: Effect of Processing Temperature on Iron Absorption From Iron Fortified Rice in Young Women
Brief Title: Iron Absorption From Fortified Extruded Rice Using Different Extruding Temperatures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Iron_ExtrudedRice
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Iron-deficiency
Keywords: Iron deficiency; iron fortified rice; extruded rice
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Reference meal (Active Comparator): 50 g of Commercial Rice was cooked and 4 mg iron from Ferrous sulphate was added Prior to give to participants. Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Reference meal
- Test meal A (Experimental): Commercial Rice was mixed with cold-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal A
- Test meal B (Active Comparator): Commercial Rice was mixed with warm-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal B
- Test meal C (Experimental): Commercial Rice was mixed with hot-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal C
- Test meal D (Experimental): Commercial Rice was mixed with cold-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal D
- Test meal E (Active Comparator): Commercial Rice was mixed with warm-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal E
- Test meal F (Active Comparator): Commercial Rice was mixed with hot-extruded fortified Rice (mixing Ratio: 100:1) Rice meal consumed with mixed vegetable Sauce.
  Interventions: Dietary Supplement: Test meal F

INTERVENTIONS:
Dietary Supplement: Reference meal — 50 g of Commercial Rice (Jasmin Rice) (dry weight) was cooked and 4 mg iron from Ferrous sulphate was added Prior to give to participants. Rice meal consumed with mixed vegetable Sauce.
  Arms: Reference meal
Dietary Supplement: Test meal A — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate, Rice meal consumed with mixed vegetable Sauce.
  Cold temperature extruding process (30-40 C°) was used to produce the extruded rice.
  Arms: Test meal A
Dietary Supplement: Test meal B — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate, Rice meal consumed with mixed vegetable Sauce.
  Warm temperature extruding process (60-70 C°) was used to produce the extruded rice
  Arms: Test meal B
Dietary Supplement: Test meal C — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate, Rice meal consumed with mixed vegetable Sauce.
  Hot temperature extruding process (80-100 °C) was used to produce the extruded rice.
  Arms: Test meal C
Dietary Supplement: Test meal D — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate,citric acid and trisodium Citrate. Rice meal consumed with mixed vegetable Sauce.
  Cold temperature extruding process (30-40 C°) was used to produce the extruded rice.
  Arms: Test meal D
Dietary Supplement: Test meal E — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate,citric acid and trisodium Citrate. Rice meal consumed with mixed vegetable Sauce.
  warm temperature extruding process (60-70 C°) was used to produce the extruded rice.
  Arms: Test meal E
Dietary Supplement: Test meal F — Commercial Rice (Jasmin Rice) was mixed with iron fortified extruded rice co-fortified with zinc sulfate,citric acid and trisodium Citrate. Rice meal consumed with mixed vegetable Sauce.
  Hot temperature extruding process (80-100 C°) was used to produce the extruded rice.
  Arms: Test meal F

SUMMARY:
Food fortification is regarded as a safe and cost-effective approach to counteract and prevent iron deficiency. Rice is a staple food for millions of people living in regions where iron-deficiency anaemia is a significant public health problem. Therefore, rice may be a promising fortification vehicle.

Hot and cold extrusion, have been identified as the major methods for rice fortification. Extruded rice has the advantage of incorporating vitamins and minerals into the food matrix.

Cold, warm and hot extrusion differ in the processing temperature and the physical structure of fortified rice kernel matrix. A recent human study in young women showed fractional iron absorption was higher in cold extruded rice compared to hot extruded Rice and this was associated with changes in the starch microstructure. These changes cannot be detected in warm extruded rice, thus, our aim is to test the iron bioavailability in difference extrusion methods; hot and warm and cold with and without the solubilizing agent CA/TSC. This will provide information on optimized rice formulations for optimal iron delivery.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years old
* Normal body Mass Index (18.5 - 25 kg/m2)
* Body weight ≤ 65 kg
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by self-declaration)
* Lactating up to 6 weeks before study initiation
* Anaemia (Hb < 12.0 g/dL)
* Elevate CRP (>5.0 mg/L)
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using Fe stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments)
* Smokers (> 1 cigarette per week)
* Difficulties with blood sampling
* Male gender
* Do not understand English

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 6 in the isotopic ratio of iron in blood at week 8 | 6 weeks, 8 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 8 in the isotopic ratio of iron in blood at week 10 | 8 weeks, 10 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
Haemoglobin | 2, 4,6,8 and 10 weeks
  Haemoglobin of each timepoint
Plasma Ferritin | 2, 4, 6, 8 and 10 weeks
  Plasma Ferritin of each timepoint
Inflammation marker | 2, 4, 6, 8 and 10 weeks
  Plasma Ferririn of each timepoint

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Scheuchzer P, Zimmerman MB, Zeder C, Sanchez-Ferrer A, Moretti D. Higher Extrusion Temperature Induces Greater Formation of Less Digestible Type V and Retrograded Starch in Iron-Fortified Rice Grains But Does Not Affect Iron Bioavailability: Stable Isotope Studies in Young Women. J Nutr. 2022 May 5;152(5):1220-1227. doi: 10.1093/jn/nxab435. PMID 34967894